CLINICAL TRIAL: NCT04616365
Title: Planned Semi-Elective Lung Transplantation Using 10°C Cold Static Preservation: A Proof-Of-Concept Study
Brief Title: Planned Semi-Elective Lung Tx Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-6364
Record Dates: First submitted 2020-08-25; First posted 2020-11-04 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi-Elective Lung Transplantation (Experimental): Planned Semi-Elective Lung Transplantation Using 10°C Cold Static Preservation
  Interventions: Procedure: Semi-Elective Lung Transplantation

INTERVENTIONS:
Procedure: Semi-Elective Lung Transplantation — When suitable donor lungs become available for a consented recipient, the transplant procedure (anesthesia starting time) will be allowed to begin earliest at 6am with the lungs being preserved at 10°C cold static preservation upon organ arrival to our hospital using a specific incubator, regardless of when donor cross clamp occurs. The maximum time allowed between donor cross clamp and recipient anesthesia initiation will be 12h.

SUMMARY:
In the current practice of lung transplantation, transplants are performed on a 24/7 schedule with a significant amount of procedures occurring overnight in order to minimize organ ischemic time. However, transplantation during the day time may lead to several advantages related to patient safety, including the presence of rested staff performing optimally, larger number of in-house professionals for emergency situations, and professional well-being. Advances and refinements in preservation practices have evolved to show that extended periods of preservation can be achieved without compromising outcome. Based on this, it is hypothesized that the avoidance of nighttime lung transplantation through prolonged pulmonary preservation will lead to at least similar patient outcomes compared to the current practice of 24/7 transplantation. During the period of this study, overnight transplants will be moved to a later start time (earliest 6AM). If lungs meet criteria for direct transplantation, they will be preserved with cold static preservation at 10°C within a special refrigerator. The maximum preservation time from donor cold flush to recipient anesthesia start time will be 12 hours.

ELIGIBILITY:
Recipient inclusion criteria

* Primary lung transplantation
* Informed consent provided
* 18-80 years old

Recipient exclusion criteria

* Re-transplantation
* Multi-organ transplantation
* >80 years old

Donor inclusion criteria

* Age ≤70 years old
* Donor lungs are suitable to go straight to lung transplantation

Donor exclusion criteria

* Age >70 years old
* Concerns with organ preservation technique
* Donor lungs require assessment by Ex Vivo Lung Perfusion (EVLP)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-04-24 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence of ISHLT Primary Graft Dysfunction Grade 3 | 72 hours post-transplant

SECONDARY OUTCOMES:
Overall survival | 30 days, 1 year post-transplant
Time on ventilator | Perioperative
ICU and hospital length of stay | Perioperative
Occurrence of acute rejection | 1 year post-transplant
Six minute walk test | 1 year post-transplant
Forced expiratory volume - one second (FEV1 in L) | 1 year post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Cypel, MD MSc, Principal Investigator — University Health Network, Toronto
Locations (3):
- Medical University of Vienna, Vienna, Austria
- University Health Network (Toronto General Hospital), Toronto, Ontario, Canada
- Hospital Universitario Puerta de Hierro-Majadahonda, Madrid, Spain

REFERENCES:
- [Derived] Iskender I. Technical Advances Targeting Multiday Preservation of Isolated Ex Vivo Lung Perfusion. Transplantation. 2024 Jun 1;108(6):1319-1332. doi: 10.1097/TP.0000000000004992. Epub 2024 May 23. PMID 38499501
- [Derived] Ali A, Hoetzenecker K, Luis Campo-Canaveral de la Cruz J, Schwarz S, Barturen MG, Tomlinson G, Yeung J, Donahoe L, Yasufuku K, Pierre A, de Perrot M, Waddell TK, Keshavjee S, Cypel M. Extension of Cold Static Donor Lung Preservation at 10 degrees C. NEJM Evid. 2023 Jun;2(6):EVIDoa2300008. doi: 10.1056/EVIDoa2300008. Epub 2023 Apr 20. PMID 38320127